CLINICAL TRIAL: NCT06026475
Title: Role of Goal Directed Fluid Therapy in Enhanced Recovery After Surgery in Gastro-intestinal Onco-surgeries
Brief Title: Role of Goal Directed Fluid Therapy in Enhanced Recovery After Surgery in Gastro-intestinal Oncosurgeries
Acronym: GDFT ERAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr Anita Kulkarni, Principal Investigator, Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RGCIRC-GDFT
Record Dates: First submitted 2023-07-29; First posted 2023-09-07 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Fluid Loss; Enhanced Recovery
Keywords: Goal Directed Fluid Therapy; Stroke volume variation; Enhanced recovery after surgery

STUDY DESIGN:
Intervention Model Description: Patients in Conventional Group will be given intraoperative fluids guided by CVP Values .
  Patients in GDFT Group will be given fluids guided by SVV values.
Who Masked: Participant
Masking Description: Participant will be masked about allotment of interventional group either CVP or SVV .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoperative Goal Directed Fluid Therapy (GDFT) guided by Stroke Volume Variation (SVV) (Active Comparator): When SVV values will increase above 11 colloid bolus 200ml will be administered. postbolus change in values of SVV , SV , SVI and CI shall be noted.
  Interventions: Procedure: Goal directed Fluid Therapy
- Intraoperative Conventional Fluid Therapy (CFT) guided by Central Venous Pressure (CVP) . (Active Comparator): When CVP values will decrease below 8 cmsH20 colloid bolus 200ml will be administered .Postbolus change in values shall be noted .
  Interventions: Procedure: Conventional Fluid Therapy

INTERVENTIONS:
Procedure: Goal directed Fluid Therapy — Patients will receive fluid during surgery with goal of maintaining SVV below 11
  Arms: Intraoperative Goal Directed Fluid Therapy (GDFT) guided by Stroke Volume Variation (SVV)
Procedure: Conventional Fluid Therapy — Patients will receive fluid during surgery with goal of maintaining CVP between 8-12 cms H20
  Arms: Intraoperative Conventional Fluid Therapy (CFT) guided by Central Venous Pressure (CVP) .

SUMMARY:
Enhanced recovery after surgery (ERAS) protocols are multimodal perioperative care pathways designed to achieve early recovery and reducing postoperative morbidity after surgical procedures by maintaining preoperative organ function and reducing the profound stress response following surgery .The key elements of ERAS protocols include preoperative counselling, optimization of nutrition, standardized analgesic and anesthetic regimens , goal directed fluid therapy early mobilization.

DETAILED DESCRIPTION:
For the proposed study investigators plan to include total 60 patients with 30 each allotted to GDFT(SVV) and CVP Group ,belonging to ASA ( American Society of Anesthesiology)Grade I/II/III, study will be conducted after obtaining written informed consent from all patients and approval from the scientific committee and Institutional Review Board (IRB). All patients will receive one-third starvation fluid as crystalloid during first hour of surgery . Night prior to and on the day of surgery carbo load will be given to all patients according to the protocol.Monitoring included 5 lead ECG SPO2,ETCO2, Invasive Blood Pressure (IBP - Radial),CVP(site IJV),core Temperature .

Standard General anaesthesia with oral Endotracheal tube and Intermittent Positive Pressure Ventilation will be given to all patients.Patients will be allotted randomly to either Goal Directed Fluid Therapy (GDFT) /SVV - Stroke Volume Variation or Conventional Central Venous Pressure - CVP guided fluid Therapy Group.

During the surgery - Heart rate , Mean arterial Blood Pressure , Urine output , Blood loss , Seum lactate levels will be noted.

For SVV Group - SVV , Stroke Volume Index (SVI) , Systemic vascular resistance index (SVRI) ,Cardiac Index (CI) values will be noted every 30 minutes- the goal is to maintain SVV value >11 and to give colloid bolus 200ml whenever SVV values rise above11.Pre and post bolus SVV, SV, SVI and SVRI shall be recorded.

For CVP Group - Goal is to maintain CVP values between 8-12 cmsH20 and for decrease in value < 8 colloid bolus of 200ml will be given and change in CVP value will be noted.

Patients in both the groups will receive Noradrenaline infusion if MAP <70 mmHg with optimal fluid transfusion .Target for transfusing Packed red blood cells will be value of haematocrit < 24 Postoperative HR, MAP, I/O-charting, Serum Creatinine, Serum Lactate, bowel sounds, Inotrope requirement, Visual Analogue Score, Ryles Tube Feeds, Epidural analgesia ,Length of stay (hours in SICU) and any postoperative complications shall be noted.

ELIGIBILITY:
Inclusion Criteria:

* Elective major open gastrointestinal Oncosurgeries .

Exclusion Criteria:

* Patient refusal.
* Robotic surgery.
* Laparoscopic surgery.
* Arrythmias.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Duration of ICU stay | upto 5 days .
  Time of shifting of patients in both group to the ward in hours.
Postoperative serum Lactate levels mmol/L | upto 48 hours
  Serum lactate levels will be measured in the SICU

SECONDARY OUTCOMES:
Serum Creatinine levels mg/dL. | Upto 48 hours.
  Serum Creatinine levels will be measured in the SICU .

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kulkarni, MD, Principal Investigator — Rajiv Gandhi Cancer Institute and Research Centre , Delhi , India
Locations (1):
- Anita Kulkarni, New Delhi, Please Select, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chong MA, Wang Y, Berbenetz NM, McConachie I. Does goal-directed haemodynamic and fluid therapy improve peri-operative outcomes?: A systematic review and meta-analysis. Eur J Anaesthesiol. 2018 Jul;35(7):469-483. doi: 10.1097/EJA.0000000000000778. PMID 29369117